CLINICAL TRIAL: NCT03026387
Title: Evaluation of the Risk Associated With Impulsivity and Other Neuropsychological Factors on Suicidal Relapse Within Hospital Emergencies
Acronym: SUI-PREDICT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: National Institute of Health and Medical Research 1061, Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UF 9681; 2016-A00845-46 (Other: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Suicide Attempt
Keywords: Suicidal behavior; Suicide attempt; Emergency department; Psychometrics; Neuropsychological tests; Suicidal ideation
MeSH Terms: conditions — Suicide, Attempted; Emergencies; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuropsychological battery tests (Other): All participants performed the same evaluation: clinical and neuropsychological assessment.
  All of them are suicide attempters without psychotic features
  Interventions: Behavioral: Neuropsychological battery tests

INTERVENTIONS:
Behavioral: Neuropsychological battery tests — The neuropsychological battery tests is composed with: Continuous Performance Test, Iowa Gambling Test, Verbal fluency (animals), Emotional stroop, Self-injury implicit association test and N-back test.
  The neuropsychological battery assesses domains heavily involved in suicidal behavior: impulsivity, affective dysregulation, alterations in decision-making (risky choices), selective attention,verbal fluidity and working memory.

SUMMARY:
Suicidal behavior (SB) is a major public health problem in France, with over 10,000 suicides (6th in the EU28) and 220,000 suicide attempts (SA) per year. These data seem underestimated by 20%. A large percentage of men (6%) and women (9%) in France made at least one lifetime SA. In addition, SBs are common among young people and are the second leading cause of death among 15-44 year-olds. The interaction of multiple factors in SB complicates the creation of predictive models. These are currently imprecise and prevent the development of consensual recommendations for the management of suicidal patients.

Most suicide attempters are evaluated in the emergency room where it is imperative to identify people with a high risk of relapse. Risk assessment is generally based on the experience of the practitioner who uses psychometric scales as support for clinical decisions. This assessment could be improved and supplemented by other sources of information. Thus, we aim to develop a short and specific tool that combines:

1. Neurocognitive measures carried out using computer software on domains strongly associated with SB: impulsivity, affective dysregulation, alterations in decision-making (risky choices), selective attention and verbal fluency.
2. Clinical and psychological assessment including the most predictive items of future SA: life events (environment) and personality traits (vulnerability). Suicide attempters will be assessed for SB and suicidal ideation in the emergency department. These measures will be repeated during a 12-month follow-up. We will use the data obtained to provide a more accurate measure of risk.

DETAILED DESCRIPTION:
Over 65 months, 5 emergency departments (Montpellier, Nimes, Uzès, Nice, Marseille) will recruit a total of 650 patients who attempted suicide.

* First visit: clinical and neuropsychological assessment
* Second and third visits at 6 and 12 months: assessment of SBs and suicidal relapse, clinical and neuropsychological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Have committed a suicide attempt within 7 days prior to inclusion
* Receive minimal treatment (assessed by the clinician)
* Sign the informed consent
* Be able to understand the nature, the aims and the methodology of the study

Exclusion Criteria:

* Patient with an actual or past history of psychotic disorder
* Patient not affiliated to a French social security system.
* Patient deprived of liberty (judicial or administrative decision)
* Patient aged 65 years or older with an MMSE score <24 at baseline.
* Patient in exclusion period after participation in another project
* Patient who has already achieved 4500€ of annual research allowances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of suicidal relapse according to aggressive impulsivity. | 12 months
  aggressive impulsivity will be assessed by the capacity to inhibit responses during a Continuous Performance Task (CPT)

SECONDARY OUTCOMES:
Score of a short scale of suicidal risk assessment | 12 months
  We aim to identify predictive factors of the occurrence of suicidal behavior in a non-psychotic suicidal population, in order to develop a battery of short-term tests applicable to emergencies. This short term tests will allow to establish a multidimensional score for the prediction of the risk of relapse.
Intensity of suicidal ideation assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) | 12 months
  We aim to identify predictive factors of the occurrence of suicidal behavior in a non-psychotic suicidal population, in order to develop a battery of short-term tests applicable to emergencies. This short term tests will allow to establish a multidimensional score for the prediction of the risk of relapse
Characteristics of suicidal behaviors assessed by Columbia Suicide History Form and the Columbia Suicide Severity Rating Scale | 12 months
  We aim to identify predictive factors of the occurrence of suicidal behavior in a non-psychotic suicidal population, in order to develop a battery of short-term tests applicable to emergencies. This short term tests will allow to establish a multidimensional score for the prediction of the risk of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Jorge LOPEZ-CASTROMAN, MD, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No